CLINICAL TRIAL: NCT02406040
Title: Effects of Short-term Energy Deficit on Muscle Protein Turnover
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Stuart M. Phillips, Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: not assigned
Record Dates: First submitted 2015-03-28; First posted 2015-04-01 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Obesity
Keywords: Protein synthesis; Protein breakdown; Muscle; Energy restriction
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Protein (Experimental): 2.4g protein/kg/d. The macronutrient composition will be 50:15:35 (carbohydrates:fat:protein) during Energy Restriction
  Interventions: Other: Energy Restriction
- Adequate Protein (Experimental): 1.2g protein/kg/d. The macronutrient composition will be 50:35:15 (carbohydrates:fat:protein) during Energy Restriction
  Interventions: Other: Energy Restriction

INTERVENTIONS:
Other: Energy Restriction — All meals will be provided for the duration of the energy restriction intervention and the energy deficit will be calculated based on estimated energy requirements by indirect calorimetry to provide 60% of energy requirements. In addition, one leg will be assigned to perform resistance exercise for 5 days during the 10 day energy deficit.

SUMMARY:
Weight loss through energy restriction results in the loss of both fat and muscle mass. Muscle mass is important for mobility, strength, glucose control and energy expenditure, and therefore the retention of muscle mass during energy restriction is an important goal. The retention of muscle mass depends on the balance between muscle protein synthesis (MPS) and muscle protein breakdown (MPB). It is well known that MPS is reduced during weight loss, however the effect of weight loss on MPB is currently a topic of debate. The purpose of this study is to assess the effect of short-term (10 day) weight loss (40% energy deficit) on both MPS and MPB in order to gain insight into the mechanisms causing muscle loss during energy restriction. In addition, the effect of resistance exercise and protein (both known to preserve muscle mass) on MPS and MPB will be examined

DETAILED DESCRIPTION:
An undesirable consequence of energy restriction is the loss of muscle mass. Muscle mass is determined by the the rates of two processes: muscle protein synthesis and muscle protein breakdown. It has been consistently shown that a reduced rate of muscle protein synthesis exists during energy restriction. However, it is currently unclear whether an increase in muscle protein breakdown also contributes to muscle mass loss. In addition, the effect of high protein diets and resistance exercise on muscle protein turnover during energy restriction, two interventions known to preserve muscle, remains to be investigated.We aim to demonstrate that the decrease in muscle protein synthesis is the main contributor to a negative protein balance during energy restriction. In addition, we hope to show that a higher-protein diet (2.4g/kg/d versus 1.2g/kg/d) and the addition of resistance exercise can help to maintain the muscle protein synthesis rate and thereby improve negative protein balance.The present study will be designed as a parallel group randomized controlled trial. Subjects will be given pre-packaged diets (Copper County Foods) to consume which will put them in a relative energy deficit of 40% per day. Based on random assignment, these subjects will either consume an adequate protein diet (1.2g/kg/d) or a high protein diet (2.4g/kg/d) for 10 consecutive days. Participants in the adequate protein diet will consume a ratio of 50:35:15 (carbohydrates:fat:protein) while subjects within the high protein diet will consume a ratio of 50:15:35 (carbohydrates:fat:protein). Subjects will undergo testing at baseline and following a 10 day dietary and unilateral resistance exercise intervention. Testing will consist of muscle and blood samples. Muscle protein synthesis and muscle protein breakdown will be measured using stable isotope tracers that are orally ingested (deuterated water) or infused into an antecubital vein (labelled phenylalanine tracers) before and after the 10 day diet.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 20 and 30 years inclusive
* Have a BMI between 25 and 33 inclusive

Exclusion Criteria:

* Have a body mass index less than 25 kg/m2 or greater than 33 kg/m2.
* Vegan
* History of allergy, sensitivity, or strong dislike towards dairy protein
* Smoker or user of tobacco products
* High physical activity
* Have health problems such as: renal or gastrointestinal disorders, metabolic disease, heart disease, vascular disease, rheumatoid arthritis, diabetes, poor lung function, uncontrolled blood pressure, dizziness, thyroid problems, or any other health conditions for which volunteers are being treated that might put them at risk for this study.
* Taking anti-diabetic, anti-inflammatory, platelet inhibitor, or anti-coagulant medications
* Use of an investigational drug product within the last 30 days
* Have participated in an infusion protocol in the last year
* Do not understand English or have a condition the PI believes would interfere with the ability to provide informed consent, comply with the study protocol, or which might confound the interpretation of the study results or put volunteers at undue risk

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Muscle protein turnover | Baseline and 10 days
  Change in muscle protein synthesis and muscle protein breakdown before and after the weight loss diet will be assessed. The relationship between high protein diets (parallel groups) and exercise (unilateral resistance exercise) on muscle protein turnover will also be examined. Muscle protein synthesis and muscle protein breakdown will be measured with stable isotope infusions of labelled phenylalanine tracers before and after the 10 day diet. In addition, long term muscle protein synthesis will be measured with orally ingested deuterated water.

SECONDARY OUTCOMES:
Molecular markers | Baseline and 10 days
  Change in the the transcriptional expression of genes involved in the ubiquitin-proteasome pathway (main regulator of muscle protein breakdown) measured in muscle samples obtained at baseline and following the 10 day dietary intervention by quantitative polymerase chain reaction (qPCR). These same samples will be analyzed by western blot for the expression of active and inactive isoforms of caspase-3, an important component of muscle protein breakdown. Finally, immunoprecipitation and western blot will be used to examine the ubiquitination of translation initiation factors at baseline and following the 10 day intervention

CONTACTS AND LOCATIONS:
Overall Officials: Stuart M Phillips, PhD, Principal Investigator — McMaster University
Locations (1):
- Exercise Metabolism Research Laboratory, McMaster Univeristy, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Pasiakos SM, Cao JJ, Margolis LM, Sauter ER, Whigham LD, McClung JP, Rood JC, Carbone JW, Combs GF Jr, Young AJ. Effects of high-protein diets on fat-free mass and muscle protein synthesis following weight loss: a randomized controlled trial. FASEB J. 2013 Sep;27(9):3837-47. doi: 10.1096/fj.13-230227. Epub 2013 Jun 5. PMID 23739654
- [Background] Pasiakos SM, Vislocky LM, Carbone JW, Altieri N, Konopelski K, Freake HC, Anderson JM, Ferrando AA, Wolfe RR, Rodriguez NR. Acute energy deprivation affects skeletal muscle protein synthesis and associated intracellular signaling proteins in physically active adults. J Nutr. 2010 Apr;140(4):745-51. doi: 10.3945/jn.109.118372. Epub 2010 Feb 17. PMID 20164371
- [Background] Areta JL, Burke LM, Camera DM, West DW, Crawshay S, Moore DR, Stellingwerff T, Phillips SM, Hawley JA, Coffey VG. Reduced resting skeletal muscle protein synthesis is rescued by resistance exercise and protein ingestion following short-term energy deficit. Am J Physiol Endocrinol Metab. 2014 Apr 15;306(8):E989-97. doi: 10.1152/ajpendo.00590.2013. Epub 2014 Mar 4. PMID 24595305
- [Background] Hector AJ, Marcotte GR, Churchward-Venne TA, Murphy CH, Breen L, von Allmen M, Baker SK, Phillips SM. Whey protein supplementation preserves postprandial myofibrillar protein synthesis during short-term energy restriction in overweight and obese adults. J Nutr. 2015 Feb;145(2):246-52. doi: 10.3945/jn.114.200832. Epub 2014 Dec 17. PMID 25644344